CLINICAL TRIAL: NCT01550861
Title: In Vitro Maturation (IVM) of Human Oocytes
Acronym: IVM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1201012117
Record Dates: First submitted 2012-02-16; First posted 2012-03-12 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Infertility
Keywords: infertility; in vitro maturation (IVM); in vitro fertilization (IVF); natural cycle
MeSH Terms: conditions — Infertility | interventions — In Vitro Oocyte Maturation Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In vitro Maturation (Experimental): in vitro maturation of immature oocytes
  Interventions: Procedure: in vitro maturation; Procedure: Polar Body Biopsy with preimplantation genetic screening

INTERVENTIONS:
Procedure: in vitro maturation — Maturation of immature oocytes in the laboratory following oocyte retrieval
Procedure: Polar Body Biopsy with preimplantation genetic screening — Polar body biopsy is performed on the day that the oocyte is retrieved. Microarray analysis will will be performed and compared with FISH and microarray analysis of day 3 or day 5 biopsy.

SUMMARY:
The objectives of this study are to evaluate the clinical efficacy of Natural in vitro Fertilization and in vitro maturation.

DETAILED DESCRIPTION:
Collection of one mature egg from a follicle in the ovary without gonadotropin medications (natural cycle IVF) results in low pregnancy rates. One way to improve natural cycle IVF is to combine this procedure with the removal of immature eggs from the ovary and mature these eggs in the laboratory ( in vitro maturation-IVM). The in vitro mature eggs are fertilized and the resultant embryos are cultured using conventional IVF techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must be female.
2. Each subject must have an indication for COH and IVF with or without ICSI.
3. Each subject must be willing and able to provide written informed consent for the trial
4. Each subject must be 25 to ≤42 years of age at the time of signing informed consent.
5. Each subject must have a normal cervical smear result (no atypical or abnormal cells, or in case of atypical squamous or glandular cells, no signs of malignancy; corresponding to Papanicolaou [PAP] I or II) obtained within 12 months prior to signing informed consent must be available

Exclusion Criteria:

1. Subject with premature ovarian failure
2. Subject with endocrine abnormalities such as hyperprolactinaemia or thyroid dysfunction
3. Subject with malformation or absence of uterus
4. Subject has tested positive for Human Immunodeficiency Virus (HIV) or Hepatitis B (by local laboratory; results obtained within 1 year prior to signing ICF are considered valid).
5. Subject with contraindication or allergy/hypersensitivity to hCG, estrogen and progesterone

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
number of oocytes retrieved and embryos generated | 1 year

SECONDARY OUTCOMES:
live birth rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zev Rosenwaks, MD, Principal Investigator — Weill Cornell
Locations (1):
- Center for Reproductive Medicine- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: Center for Reproductive Medicine- Weill Cornell Medical College — http://ivf.org